CLINICAL TRIAL: NCT05214027
Title: The Effect of an Acute Bout of Exercise on Serum Vitamin D Concentration
Status: Completed | Type: Observational
Sponsor: University of Bath (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Sophie Davies, PhD Student, University of Bath
Other Study IDs: EP 19/20 026
Record Dates: First submitted 2022-01-12; First posted 2022-01-28 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Vitamin D; Acute Exercise
Keywords: Vitamin D; Acute Exercise; Adults; United Kingdom; Lipid Mobilisation
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Human Plasma and Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: This study follows a randomised crossover design. All participants will undergo a single 60-minute treadmill-based exercise intervention, and a resting period for equal duration in a randomised order.
  Interventions: Other: Treadmill-Based Exercise (60% VO2 Max for 60 minutes); Other: Rest (60 minutes)

INTERVENTIONS:
Other: Treadmill-Based Exercise (60% VO2 Max for 60 minutes) — Each participant will undergo a single 60-minute treadmill-based exercise intervention in a randomised order.
  Treadmill settings are generated based on settings which correspond to participants exercising at 60% VO2 max from their maximal exercise test on visit 2. To confirm that participants are exercising at 60% during the hour session, 1 minute samples of expired air are taken at 15 minute intervals and immediately analysed to check % VO2 max. Participants heart rate and RPE measures are also taken at 15 minute intervals throughout the exercise session and cross-checked against predicted values at 60% VO2 Max.
Other: Rest (60 minutes) — Each participant will undergo a 60-minute rest period in a randomised order.

SUMMARY:
Vitamin D deficiency is considered a public health priority in the UK, with approximately 30-40% of the UK population being deemed vitamin D deficient during winter months. Current government strategies to improve vitamin D status amongst the UK population involve dietary supplementation, however, it has been shown that excess adiposity reduces the impact of dietary supplementation with vitamin D. One potential explanation for this observation is that vitamin D becomes sequestered in adipose tissue. We hypothesise that exercise may facilitate the mobilisation of vitamin D from adipose tissue and thus increase circulating vitamin D (25OHD) concentrations. Little is currently known as to whether a single bout of exercise affects vitamin D status, with a handful of studies demonstrating contradictory findings. This research will examine the effect of an acute bout of exercise (treadmill-based at 60% VO2 Max for 60 minutes) on vitamin D status (serum 25(OH)D) in healthy community-dwelling adults.

DETAILED DESCRIPTION:
This study is a random crossover design and will require 34 participants to visit the University of Bath on 6 separate occasions in total.

Individuals who express an interest in taking part will be invited to attend an initial screening meeting at the University so that the eligibility can be assessed for the study, and the all procedures explained verbally. If the participant is eligible and is happy to participate in the study, they will attend a second visit prior to two trials to undertake a treadmill-based maximal exercise test (VO2 Max), resting metabolic rate measure and several measures will be taken to assess body composition. Trials will involve a 60-minute exercise bout at 60% of the participant's maximum oxygen uptake or a 60-minute resting period (both followed by a further hour of rest). The order in which these trials occur will be randomised for each participant and the participant will not be told of this order prior to the trials.

During both trials, a cannula will be inserted into a vein in the arm prior to exercise and 10ml blood samples will be drawn at baseline (pre-exercise) and immediately after the exercise session and 1 hour post exercise from the antecubital vein. The participant will return to the university the day after each trial for a 10ml venous blood sample (24hr post-exercise) which will be taken via venepuncture. In the 24 hours following a trial, participants will be provided with standardised meals in order to ensure energy balance. Other controls which will be applied during the study period will include the provision of factor 50 sunscreen (if the participant is undertaking trials between March and October) to aid in mitigating against the cutaneous synthesis of vitamin D, and guidance on avoiding any strenuous activity 24 hours prior to trial days. Participants will also be provided with a physical activity monitor (MotionWatch8, CamNTech) to wear during trial days after leaving the lab.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (see exclusion criteria)
* 25-65 years old
* Ability to travel to and from University of Bath campus

Exclusion Criteria:

* Current or recent use (within the last three months) of weight loss drugs, medication that would interfere with study outcomes, sunbeds, or dietary vitamin D supplementation
* Change in weight of more than 5% in the last six months, or a significant change in lifestyle in the last two months
* Positive responses to the Physical Activity Readiness Questionnaire (PAR-Q)
* Presence of coronary heart disease, chronic kidney disease, type 2 diabetes, stroke, heart failure, peripheral arterial disease, severe hypertension (blood pressure >180/110 mmHg)
* BMI <18kg/m2 or BMI >40kg/m2

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, community-dwelling adults (aged 25-65 years old)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D concentration | 24 hours- change from baseline to 24 hours post exercise
  As assessed by serum 25(OH)D via LC-MS

SECONDARY OUTCOMES:
Markers of lipid mobilisation | 24 hours- change from baseline to 24 hours post exercise
  As assessed by plasma NEFA, triacyglycerol and glycerol
Calcium | 24 hours- change from baseline to 24 hours post exercise
  As assessed by serum calcium
Other vitamin D metabolites | 24 hours- change from baseline to 24 hours post exercise
  As assessed by serum 1,25(OH)D and other forms of serum vitamin D via LC-MS

CONTACTS AND LOCATIONS:
Locations (1):
- Sophie Ella Davies, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No